CLINICAL TRIAL: NCT00507013
Title: The QuickClose Study: Hemostatic Closure of Femoral Artery Access Site, Using the QuickClose: a Prospective, Non-Randomized Clinical Study
Brief Title: Hemostatic Closure of Femoral Artery Access Site, Using the QuickClose
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CardioDex (Industry)
Collaborators: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RD 392-03
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Hemostasis,Surgical
Keywords: vascular closure device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Other)
  Interventions: Device: QuickClose device

INTERVENTIONS:
Device: QuickClose device

SUMMARY:
The QuickClose study is a prospective, non-randomized study, to evaluate the safety and efficacy of the QuickClose device using two different dose types of heat exposure.

Patients undergoing a diagnostic angiogram procedure will be treated with the QuickClose device. Two groups of 20 patients each, will be enrolled consecutively, Group A will complete enrollment before enrollment into Group B begins. Patients will be monitored until 30 days after the procedure

DETAILED DESCRIPTION:
The primary safety endpoint is the incidence of major complications related to method for achieving hemostasis at the puncture site. The secondary safety endpoint is the incidence of minor complications related to method for achieving hemostasis at the puncture site. The primary efficacy endpoint are time to hemostasis, time to ambulation and time to discharge . The secondary efficacy endpoints are device and procedure success.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age
2. The patient or guardian must provide written informed consent
3. The patient must be willing to comply with follow-up requirements
4. The patient has no child bearing potential or has a negative pregnancy test within the previous 7 days.
5. Patient is eligible for same day discharge

Procedural Inclusion:

1. A intravascular procedure was preformed using 6 Fr introducer
2. The introducer sheath is located in the common femoral artery

Exclusion Criteria:

1. Manual compression has been preformed on the ipsilateral arterial site within the previous 6 weeks
2. Any closure device has been used on the ipsilateral arterial site within the previous 180 days
3. Any reentry of the ipsilateral site is planned within the next 6 weeks.
4. History of surgical repair of blood vessels of the ipsilateral arterial site
5. Significant bleeding diathesis or platelet dysfunction

   1. Thrombocytopenia (Plt count ≤ 100,000)
   2. Anemia (Hgb ≤ 10mg/dl and/or Hct ≤ 30mg/dl)
6. Has life expectancy of less than 1 year due to terminal illness
7. Currently being treated for an infection
8. Receiving GP 2b/3a inhibitors or requires warfarin therapy within the last 14 days.
9. INR results > 1.2 on day of procedure
10. Experienced a Myocardial infarction (CK-MB ≥ 2x upper limits of normal) within the previous 72 hours
11. Received thrombolytic within previous 72 hours
12. Patient is currently enrolled in an investigational device or drug study which endpoints have not been met.
13. Absent of pedal pulse
14. Pre-existing autoimmune disease (i.e., Lupus, Addison's Disease, Grave's Disease)
15. Has Body Mass Index(BMI) <20, or BMI >40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
rate of complication | 30 days

SECONDARY OUTCOMES:
time to hemostasis | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Amit Segev, MD, Principal Investigator — The Chaim Sheba Medical Center
Locations (1):
- The Chaim Sheba M.C., Tel Litwinsky, Israel